CLINICAL TRIAL: NCT06855407
Title: The Effects of Induced Hypertension on Cerebrovascular Hemodynamics During General Anaesthesia
Brief Title: Hypertension and Cerebrovascular Hemodynamics in General Anaesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Region Västerbotten (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-05508-02
Record Dates: First submitted 2025-02-28; First posted 2025-03-03 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Anesthesia; Cerebral Blood Flow; Regional Cerebral Oxygen Saturation; Blood Pressure
Keywords: induced hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Change in cerebral blood flow with increased systemic blood pressure during general anesthesia (Experimental)
  Interventions: Other: Blood pressure elevation

INTERVENTIONS:
Other: Blood pressure elevation — Increasing systemic blood pressure for measurement of cerebral blood flow changes

SUMMARY:
During anesthesia, blood pressure-raising medications are often required to achieve an adequate blood pressure level. However, there is limited knowledge about what constitutes an adequate blood pressure to ensure sufficient blood flow to the brain. This project aims to map the relationship between blood pressure and brain blood flow using an MRI scanner. The results will contribute to a better understanding of this relationship and lead to improved management of brain blood flow during surgery on anesthetized patients.

How does the project work?

Day 1 Before planned surgery, participants will meet with an anesthesiologist for information and assessment. An MRI scan of the brain will be conducted while participants are awake. The MRI examination has no side effects or risks. The space inside the MRI scanner is tight, especially around the head. If discomfort is experienced, the examination will be stopped immediately. The machine is noisy, so hearing protection will be provided, and communication with staff will be possible throughout the examination. The scan takes approximately 30 minutes, during which participants only need to lie still and relax.

Day 2 After planned surgery, an anesthesiologist and an anesthesia nurse will transfer participants to the MRI scanner while still under anesthesia. Participants will not be woken up between surgery and the MRI scan; instead, transportation will occur while still anesthetized, following standard hospital procedures.

Participants will remain under the same anesthetic drugs as during the surgery. The same blood pressure-raising medication, norepinephrine, will be continuously used.

No additional drugs, beyond those necessary for normal anesthesia, will be administered before the MRI examination.

The entire project will take about 1.5 hours in addition to the surgery. If an arterial catheter (a blood pressure monitor via an artery in the wrist) is not already in place, one will be inserted while participants are asleep.

Before the MRI examination:

Baseline examination - If any abnormalities are detected, the scan will be stopped, and follow-up by a doctor will occur.

Blood pressure increase - Blood pressure will be raised by approximately 30% (equivalent to mild physical activity, such as jogging).

Follow-up scan at the higher blood pressure level. Blood pressure returns to normal. All blood pressure levels will remain within clinically acceptable ranges for anesthetized patients and will be regulated with the same medication as used during the surgery.

After the MRI:

Participants will be woken up in the anesthesia preparation room next to the MRI scanner.

The arterial catheter will be removed before awakening. Participants will be transported to the postoperative unit for monitoring. The surgeon responsible for care will determine the discharge time.

Possible Risks and Side Effects of Participation

Transporting an anesthetized patient for an MRI scan outside the operating room carries some risks. However, the hospital has established procedures for daily transportation of anesthetized patients and a structured division of responsibilities to manage unexpected situations. Monitoring will be conducted by an experienced anesthesiologist and anesthesia nurse throughout the procedure.

Routine monitoring includes blood pressure, heart rate, depth of anesthesia, and oxygen levels.

No long-term effects have been observed from MRI scans or short-term anesthesia for these examinations.

Most complications related to general anesthesia occur during induction or awakening, and these risks exist regardless of study participation.

Study participation may slightly increase the risk of IV lines or breathing tubes becoming dislodged due to movement while anesthetized.

A prolonged period under anesthesia may cause slight additional fatigue upon waking.

To ensure understanding of the information about this study, participants will take a simple cognitive test (5 minutes) before surgery.

If any unexpected complications arise during surgery, study participation will be discontinued. If the MRI scan reveals any abnormalities, referral to a neurologist or neurosurgeon for further evaluation will be provided.

What Happens to Collected Data?

The project will collect health information from medical records and MRI scans. All data will be pseudonymized (coded) so that it cannot be linked to individual participants.

The key to decoding this information will be stored securely by the research nurse at the Neuro-Head-Neck Center (NHHC).

Only authorized research personnel will have access to the pseudonymized data. Information will be protected in accordance with the General Data Protection Regulation (GDPR).

DETAILED DESCRIPTION:
The Impact of Blood Pressure on Cerebral Blood Flow: An MRI Study on Neuroprotective Blood Pressure Thresholds During Anesthesia

Abbreviations Used in the Research Program

ASA - American Society of Anesthesiologists Classification

ASL - Arterial Spin Labeling

BP - Blood Pressure

CBF - Cerebral Blood Flow

CO - Cardiac Output

CPP - Cerebral Perfusion Pressure

CVR - Cerebral Vascular Resistance

CT - Computed Tomography

HR - Heart Rate

ICP - Intracranial Pressure

MAP - Mean Arterial Pressure

MRI - Magnetic Resonance Imaging

NIRS - Near-Infrared Spectroscopy

PCMRI - Phase-Contrast Magnetic Resonance Imaging

rSO2 - Regional Cerebral Oxygen Saturation

Objective and Aims Ensuring adequate cerebral perfusion (CBF) during general anesthesia is critical for maintaining sufficient oxygenation and blood supply to the brain during surgery. This regulation is primarily achieved through blood pressure adjustments (MAP) using vasopressors to maintain adequate perfusion pressure and, consequently, sufficient CBF. However, the relationship between MAP, HR, and CBF is complex, particularly as increasing MAP often necessitates increasing vascular resistance, which may paradoxically reduce blood flow. Furthermore, the autoregulatory system complicates the relationship between CVR and cerebral blood flow. Despite these complexities, MAP is considered the most relevant surrogate marker for CBF in clinical practice. Most intraoperative scenarios target a MAP of ≥65 mmHg to ensure sufficient organ perfusion regardless of gender, age, or comorbidities.

Another commonly used surrogate marker is rSO2, measured via NIRS. Impaired CBF during anesthesia has been associated with postoperative cognitive decline and confusion. To mitigate postoperative hypoperfusion-related symptoms, it is essential to determine the optimal intraoperative blood pressure management for each patient. This necessitates further research into how blood pressure regulation via commonly used anesthetic agents affects CBF.

Our hypothesis is that CBF during anesthesia and blood pressure regulation via vasopressors does not correlate with current clinical practice. This is due to significant inter-individual variations and other physiological factors, such as HR, vascular tone, and arterial pulsations, which may influence the relationship between blood pressure and cerebral blood flow. Additionally, advanced MRI techniques could facilitate a more precise understanding of the MAP-CBF relationship, leading to the development of more robust surrogate markers.

The objective of this study is to investigate the impact of blood pressure alterations using norepinephrine on cerebral hemodynamics in anesthetized subjects. This will be achieved by directly measuring MAP, HR, CO, CBF, and regional cerebral oxygenation simultaneously, a methodology not previously implemented.

Research Questions

Investigate how pharmacologically induced blood pressure elevation (20-30% above baseline) via norepinephrine affects cerebral blood flow.

Clarify the relationships among CVR, CO, MAP, HR, and CBF.

Develop a novel relationship curve between MAP and CBF.

Assess regional cerebral oxygen saturation (rSO2) via NIRS in relation to CBF using MRI under varying MAP conditions.

We will employ MRI for blood flow quantification in major cerebral vessels (PCMRI) and brain tissue (ASL), while also measuring rSO2 using NIRS. A preliminary study on healthy, awake volunteers demonstrated that norepinephrine-induced MAP elevation correlates with increased CVR and reduced CO, ultimately leading to decreased CBF despite the higher MAP. These findings could significantly influence current perceptions of the MAP-CBF relationship and improve intraoperative safety by reducing the risk of postoperative complications associated with cerebral hypoperfusion.

Background and Literature Review

Cerebral Blood Flow and Systemic Blood Pressure Clinical blood pressure regulation during surgery is goal-directed, with MAP ≥65 mmHg serving as the lower threshold to prevent organ damage. CBF is closely linked to CPP, which in turn is strongly associated with MAP. In intraoperative settings, MAP can be increased either by raising systemic vascular resistance (SVR) or by increasing CO. However, an increase in MAP does not necessarily lead to increased CBF.

MAP serves as an indirect measure of CBF since direct clinical measurement of CBF is not feasible. Lassen's autoregulation model, established in the 1950s, describes a stable CBF within an MAP range of approximately 60-160 mmHg. However, factors such as age, comorbidities, vascular anatomical variations, and impaired autoregulation complicate the validity of this model.

Recent studies suggest a need for individualized blood pressure management during anesthesia. While cerebral perfusion in awake patients can be monitored via clinical examination, this becomes challenging under general anesthesia. Hemodynamic instability is common during anesthesia and is typically managed through fluid administration and vasopressor infusion. However, anesthetic agents often induce a reduction in MAP. Vasopressors increase MAP via vasoconstriction and CO modulation through alpha- and beta-adrenergic receptor activation. The optimal intraoperative MAP threshold remains uncertain, highlighting the need for a better understanding of the mechanistic interactions between MAP regulation and CBF.

Cerebral Oxygenation and Blood Flow NIRS is a non-invasive technique that uses near-infrared light (700-850 nm) to measure regional cerebral oxygen saturation (rSO2) at a depth of approximately 1.7 cm. It is increasingly utilized perioperatively for monitoring brain oxygenation and early detection of cerebral ischemia and hypoxia. However, uncertainties remain regarding the clinical impact of active cerebral NIRS monitoring on postoperative outcomes.

Methodology for Cerebral Blood Flow Measurement Previous studies on the MAP-CBF relationship relied on invasive techniques, often conducted in animal models. Recently, non-invasive methods such as NIRS and transcranial Doppler have been utilized; however, these serve as surrogate measures of blood flow and carry a high risk of misinterpretation. PCMRI is the only current non-invasive technique that provides absolute CBF measurements. At Umeå University, PCMRI is an established method for studying cerebral hemodynamics and is considered the gold standard for non-invasive blood flow measurement. Combining PCMRI and ASL with invasive blood pressure monitoring allows for a comprehensive assessment of the relationship between cerebral blood flow, perfusion, and systemic blood pressure.

Knowledge Gaps The established understanding of the MAP-CBF relationship is frequently questioned, with no widely accepted alternative models for clinical application. Current blood pressure thresholds in anesthesia are generalized rather than patient-specific and do not account for physiological parameters or the method used to achieve target values. Many studies underpinning clinical practice are outdated, based on indirect measurement methods, or conducted in animal models. The use of surrogate markers for intraoperative cerebral perfusion remains limited, as their direct correlation with postoperative outcomes is unclear. This necessitates simultaneous measurements of relevant physiological parameters using reliable direct methods.

Clinical Significance Cognitive impairment, delayed recovery, and increased mortality have been linked to inadequate cerebral perfusion during anesthesia and intensive care. This not only affects patient well-being but also increases healthcare costs and length of hospital stay. A robust, individualized hemodynamic parameter strongly associated with CBF is necessary. If pharmacologically controlled blood pressure does not align with current knowledge of its effects on cerebral blood flow, its role in anesthesia should be re-evaluated. Additionally, rSO2 measured via NIRS should be further investigated due to its potential for seamless integration into clinical practice.

This project, with strong clinical implications, also incorporates a physiological research component to better understand the interplay of various physiological factors. By employing direct methods to measure CBF and obtain absolute values, we aim to generate robust data to redefine the MAP-CBF relationship and assess whether current intraoperative blood pressure management is beneficial for patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification 1-3
* BMI 18,5-29.9
* MMSE > 23
* Elective surgery planned.

Exclusion Criteria:

- Pacemaker or other contraindications for MRI.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2026-12-06 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Cerebral blood flow | 1 hour
  mL/min as measured by MRI
rSO2 | 1 hour
  Regional oxygen saturation index

CONTACTS AND LOCATIONS:
Locations (1):
- Umeå University Hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Osterlind J, Birnefeld J, Birnefeld E, Hultin M, Qvarlander S, Wahlin A, Holmlund P, Zarrinkoob L. Study protocol: MRI-based assessment of cerebral blood flow under pharmacologically elevated blood pressure in patients under general anesthesia, and in sedated ICU patients with aneurysmal subarachnoid hemorrhage. PLoS One. 2025 Dec 10;20(12):e0338688. doi: 10.1371/journal.pone.0338688. eCollection 2025. PMID 41370289